CLINICAL TRIAL: NCT06804928
Title: Investigation of the Effect of Virtual Reality Glasses Used During Extracorporeal Shock Wave Lithotripsy (ESWL) on Patients' Pain, Anxiety, and Comfort Levels: A Randomized Controlled
Brief Title: Effect of Virtual Reality Glasses on Pain, Anxiety, and Comfort During Extracorporeal Shock Wave Lithotripsy
Acronym: ESWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Seda Cansu Yeniğün, Lecturer Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Scansuscansu92
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: ESWL; Anxiety; Pain; Comfort; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The measurements will be conducted by an individual independent of the study. Additionally, the statistical analysis of the research will be performed by a statistician who is unaware of the study details. The randomization plan was also prepared by a researcher independent of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-G (Virtual Reality Group) (1) (Experimental): During the procedure, the patient will wear virtual reality glasses and watch a video. The video will be played through the virtual reality glasses throughout the entire procedure.
  Interventions: Behavioral: Virtual Reality Glasses
- Control Group (2) (No Intervention): No intervention will be applied to the patients in the control group, and the standard care protocol of the clinic will be followed.

INTERVENTIONS:
Behavioral: Virtual Reality Glasses — During the procedure, the patient will wear virtual reality glasses and watch a video. The video will be played through the virtual reality glasses throughout the entire procedure.
  Other Names: Control group
  Arms: VR-G (Virtual Reality Group) (1)

SUMMARY:
Effect of Virtual Reality Glasses on Pain, Anxiety, and Comfort During ESWL

ELIGIBILITY:
Inclusion Criteria:

Being 18 years of age or older, Having no hearing or perception impairments, Having no visual impairments, Undergoing ESWL for the first time.

Exclusion Criteria:

Use of any analgesic or anxiolytic medication before the procedure, Having a psychiatric disorder, The procedure being performed on an emergency basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
VAS | Data will be collected 10 minutes before the procedure.
  Pain levels will be assessed.
Visual Anxiety Scale (VAS-A) | Data will be collected 10 minutes before the procedure.
  Anxiety levels will be assessed.
Visual Comfort Scale | Data will be collected 10 minutes before the procedure.
  Comfort levels will be assessed.
Spielberger Trait Anxiety Inventory (STAI-II) | The measurement will be conducted only once, 10 minutes before the procedure.
  It will be used to measure trait anxiety levels before the procedure.
VAS | Data will be collected 30 minutes after the procedure.
  Pain levels will be assessed.
Visual Anxiety Scale (VAS-A) | Data will be collected 30 minutes after the procedure.
  Anxiety levels will be assessed.
Visual Comfort Scale | Data will be collected 30 minutes after the procedure.
  Comfort levels will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun Gazi State Hospital, Samsun, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided